CLINICAL TRIAL: NCT04657146
Title: Longitudinal Assessment of Marrow and Blood in Patients With Glioblastoma
Acronym: LAMB-G
Status: Suspended | Type: Observational
Why Stopped: Study undergoing amendment and funding changes.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107040
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma
Keywords: Glioblastoma, T cells, Sequestration; Sphingosine-1-phosphate receptor 1; β-arrestin, Bone marrow, Immunotherapy
MeSH Terms: conditions — Glioblastoma | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Tumor collection
  2. Peripheral blood sample collection
  3. Bone marrow aspiration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected newly-diagnosed Glioblastoma (GBM): Patients, ≥18 years of age, with newly diagnosed GBM, World Health Organization (WHO) Grade IV, undergoing gross total resection (defined as >90% of contrast enhancing volume removed on post-operative MRI) and collection of blood, bone marrow, and tumor.
  Interventions: Other: Biorepository

INTERVENTIONS:
Other: Biorepository — Tumor collection (> 1cm3): Intraoperatively
  Peripheral blood collection:
  * Intraoperatively (60mL +/- 5mL)
  * Post-resection (30mL +/- 5mL)
  * Post- standard of care treatment (30mL +/- 5 mL)
  Bone marrow aspiration:
  * Intraoperatively (10mL +/- 5 mL)
  * Post-resection (5mL +/- 5 mL)
  * Post- standard of care treatment (5mL +/- 5 mL)

SUMMARY:
The main goal of this study is to provide foundational data to drive translational approaches for an entirely novel category of immunotherapy.

DETAILED DESCRIPTION:
The investigators' recent studies show that large numbers of T cells in patients and mice with intracranial tumors are sequestered in bone marrow. This phenomenon mysteriously confines a pool of functional, naïve T cells with anti-tumor capacity to a compartment where they are unable to access tumor, eliciting a mode of T cell dysfunction categorized as "ignorance." The investigators have uncovered that loss of the sphingosine-1-phosphate receptor 1 (S1P1) from the surface of T cells mediates their sequestration in bone marrow, while blocking internalization of S1P1 facilitates stabilization of the receptor on T cells and frees them for anti-tumor activities. As the investigators look to design interventions targeting β-arrestin mediated S1P1 internalization as a novel anti-tumor strategy, they need to better understand variations in sequestration across patients, over time, and with treatment. Assessing these variations and biomarkers that may accompany them will help to establish a target treatment population, as well as the optimal timing for intervention.

Primary Objectives:

1. Assess variations in blood and bone marrow T cell counts as they relate to treatment time-points in patients with glioblastoma (GBM).
2. Assess variations in S1P1 levels and their correlation with blood and bone marrow T cell counts over the course of treatment in patients with GBM

Exploratory Objectives:

1. Assess the associations between tumor size and degree of lymphopenia and bone marrow T cell sequestration observed.
2. Compare The Cancer Genome Atlas (TCGA) subclasses with respect to the degree of lymphopenia and bone marrow T cell sequestration observed at diagnosis.
3. Examine patient plasma, tumor supernatant, and tumor ribonucleic acid (RNA) for markers that are associated with lymphopenia, T cell S1P1 levels, and bone marrow T cell sequestration. Initial candidates will include transforming growth factor-β (TGFβ) 1/2, tumor necrosis factor (TNF), interleukin (IL)-33, IL-6, catecholamines, signal transducer and activator of transcription 3 (STAT3) RNA, and Kruppel-like factor 2 (KLF2) RNA.
4. Compare T cell phenotypes in the blood and bone marrow of patients exhibiting versus not exhibiting T cell lymphopenia or sequestration.
5. Compare differences in tumor-infiltrating lymphocyte numbers and phenotypes between patients with and without lymphopenia / sequestration at diagnosis.
6. Establish baseline β-arrestin 1 and 2 expression in patients and assess variation across individuals.
7. To determine cellular component of the bone marrow upon collection of enough samples to batch. Numbers of various bone marrow resident cells will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age.
* Suspected newly-diagnosed GBM, World Health Organization (WHO) Grade IV with intent for gross total resection (as defined above).
* Accessibility for treatment and follow up.
* Patient consent obtained according to Duke institutional policy.
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test according to standard of care prior to surgery.

Exclusion Criteria:

* Patients who previously received other conventional therapeutic interventions for newly diagnosed glioblastoma with the exception of surgical intervention.
* Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Pregnant or breast-feeding during the study period.
* Patients with an active infection, or febrile within 24 hours of surgery.
* Patients with inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, or other autoimmune disease.
* Patients with history of or active hematologic or bone marrow diseases, including but not limited to diagnosed lymphomas, leukemias, sickle cell or other anemias not associated with their current condition or polycythemia vera.
* Prior bone marrow harvests preceding this study.
* Patients with known or suspected immunodeficiency or human immunodeficiency virus (HIV).
* Hematocrit < 24 % pre-operatively.
* Patients with a serious active infection or other serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment or comply with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the terms of the inclusion and exclusion criteria above will be eligible to participate in the study. This includes all patients over 18 years of age, both sexes, and all minorities. A total of 40 patients will be enrolled in the study. Patients who are not confirmed to have GBM on histopathological analysis, or who do not qualify as gross total resection per the definition above will be removed from the study and replaced until a total of 40 patients is reached.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Variations in blood and bone marrow T cell counts | 2 years
  Assess variations in blood and bone marrow T cell counts as they relate to treatment time-points in patients with glioblastoma.
Variations in Sphingosine-1-phosphate receptor 1 (S1P1) levels | 2 years
  Assess variations in S1P1 levels and their correlation with blood and bone marrow T cell counts over the course of treatment in patients with glioblastoma.

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Patel, M.D., Principal Investigator — Duke University; Katayoun Ayasoufi, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No